CLINICAL TRIAL: NCT00596440
Title: Assessment of a Teachable Moment for Smoking Cessation
Acronym: TM
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Robert Schnoll, Associate Professor, University of Pennsylvania
Other Study IDs: 805712; NIH R01CA126969
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Nicotine Dependence
Keywords: smoking; teachable moment; cancer
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Neoplasms | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Relatives of Cancer Patients
  Interventions: Drug: Transdermal nicotine patch
- 2: Relatives of Orthopedic Patients
  Interventions: Drug: Transdermal nicotine patch

INTERVENTIONS:
Drug: Transdermal nicotine patch — 8 weeks; 4 weeks of 21mg, 2 weeks of 14mg, and 2 weeks of 7mg.

SUMMARY:
A teachable moment (TM) refers to life events or transitions, such as physician visits, early detection screening feedback, pregnancy, and hospitalization for, and diagnosis of, disease, that inspire health behavior change. Despite strong intuitive appeal of the TM concept and over 150 studies of interventions implemented in a TM, there has been little investigation of the influence of TMs for smoking, particularly for promoting smoking cessation among those indirectly affected by a TM (e.g., relatives of cancer patients). This prospective observational study using a matched-group design will assess whether a lung cancer diagnosis increases enrollment in a smoking cessation program and cessation, and reduces smoking, among the patient's relatives/spouse who smoke. We will compare enrollment in a cessation program and cessation and smoking rates in 2 groups of smokers: 1) relatives/spouses of newly-diagnosed lung cancer patients, and 2) relatives/spouses of patients with an orthopedic condition. We will also explore mediators and moderators of a lung cancer diagnosis as a TM. This study could clarify the TM concept for smoking cessation, shed light on the underlying mechanisms of TMs, and guide future development and implementation of TM-based smoking cessation interventions.

ELIGIBILITY:
Inclusion Criteria:

1. A relative (i.e., sibling, parent, child, grandparent, aunt, uncle, cousin) or spouse of a newly-diagnosed lung or head and neck cancer patient or orthopedic patient (e.g., arthritis, bone and joint infection, foot and ankle conditions, hand, wrist, and elbow conditions such as carpal tunnel syndrome, shoulder and elbow conditions, such as rotator cuff injury, and knee conditions, such as ligament damage repair);
2. A regular smoker (i.e., smoke 10 cigarettes/day on average);
3. Able to use NRT (see contraindications under Key Exclusion Criteria);
4. Age 18 or older (to use NRT); and
5. Living within ~50 miles of PENN (to allow for meetings at PENN).

Exclusion Criteria:

1. Cannot communicate in English;
2. Have current alcohol abuse/dependence;
3. Are or have been diagnosed with cancer, asthma, HIV, emphysema, or COPD;
4. Have a current medical problem for which NRT is contraindicated such as uncontrolled hypertension (> 150 over 90), unstable angina, heart attack or stroke within the past 6 months, and liver and/or kidney failure in the last 6-months;
5. Currently use monoamine oxidase inhibitors or benzodiazepines, anti-psychotics, and antidepressants, including bupropion;
6. Are allergic to adhesive tape or latex, and
7. Are a female who is pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One group will be relatives/spouses of newly-diagnosed lung or head and neck cancer patients and the second group will be relatives/spouses of orthopedic patients. All participants will be regular smokers (i.e., smoke 10 cigarettes/day on average).
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2007-08; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Schnoll, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Relatives of Cancer Patients: Relatives of Cancer Patients offered Transdermal nicotine patch: 8 weeks; 4 weeks of 21mg, 2 weeks of 14mg, and 2 weeks of 7mg and behavioral counseling.
- Relatives of Orthopedic Patients: Relatives of Orthopedic Patients offered transdermal nicotine patch: 8 weeks; 4 weeks of 21mg, 2 weeks of 14mg, and 2 weeks of 7mg and behavioral counseling
Period: Overall Study
Arm/Group | Relatives of Cancer Patients | Relatives of Orthopedic Patients
Started | 113 | 121
Showed to Eligibility Visit | 85 | 72
Showed to First Treatment Session | 61 | 52
Completed | 48 | 41
Not Completed | 65 | 80

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Relatives of Cancer Patients | Relatives of Orthopedic Patients | Total
Number analyzed (Participants) | 113 | 121 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (11.7) | 49.2 (11.7) | 47.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 70 | 127
  Male | 56 | 51 | 107

OUTCOME MEASURES:

1. Primary Outcome: Accrual Rate (Eligibility Visit)
Description: Show rate to eligibility visit
Time Frame: week zero
Measure: Number; unit: participants
Arm/Group | Relatives of Cancer Patients | Relatives of Orthopedic Patients
Number analyzed (Participants) | 113 | 121
participants | 85 | 72

2. Secondary Outcome: Smoking Cessation Rate
Time Frame: week nine
Population: The 129 participants represents a subset of the sample that participated in treatment. This subset of participants includes only those who attended eligibility session and participated in the week 9 follow-up. One oncology relative became ineligible immediately following completion of this counseling session and was excluded.
Measure: Number; unit: participants
Arm/Group | Relatives of Cancer Patients | Relatives of Orthopedic Patients
Number analyzed (Participants) | 67 | 61
participants | 13 | 16

3. Secondary Outcome: Show Rate at First Treatment Session
Time Frame: week one
Population: This analysis includes only a subset of participants who had not discontinued the study by week 1.
Measure: Number; unit: participants
Arm/Group | Relatives of Cancer Patients | Relatives of Orthopedic Patients
Number analyzed (Participants) | 112 | 117
participants | 61 | 52

ADVERSE EVENTS:
Arm/Group | Relatives of Cancer Patients | Relatives of Orthopedic Patients
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/121
Other Adverse Events (participants affected / at risk) | 0/113 | 0/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes